CLINICAL TRIAL: NCT01103492
Title: Treatment of Hemorrhagic Radiation Proctitis Using the Halo System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Covidien, GI Solutions (Industry)
Responsible Party: Principal Investigator, Jeffrey Marks, MD, Principal Investigator, University Hospitals Cleveland Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-07-46
Record Dates: First submitted 2010-04-13; First posted 2010-04-14 (Estimated); Results first posted 2011-04-27 (Estimated); Last update posted 2015-01-05 (Estimated); Status verified 2014-12

CONDITIONS: Pelvic Neoplasms
Keywords: prostate cancer; endometrial cancer; radiation proctitis; pelvic radiotherapy; rectal bleeding
MeSH Terms: conditions — Pelvic Neoplasms; Prostatic Neoplasms; Endometrial Neoplasms; Gastrointestinal Hemorrhage | interventions — Blood Coagulation Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ablation catheter (Experimental): Procedure using the HALO90 Ablation catheter to heat a thin layer of rectal tissue using radiofrequency to reduce inflammation and bleeding in subjects with radiation proctitis.
  Interventions: Device: HALO90 Ablation catheter

INTERVENTIONS:
Device: HALO90 Ablation catheter — FDA approved endoscopic device for use in coagulation of tissue in the digestive tract using radiofrequency energy.
  Other Names: Coagulation; Endoscopic Device

SUMMARY:
This study involves evaluating a procedure in which the study device, the HALO90 Ablation catheter, is used to heat a thin layer of tissue lining the rectum using radiofrequency (RF) energy in subjects suffering from radiation proctitis (acute inflammation of the inner lining of the rectum caused by the side effects of radiation treatments that can lead to bleeding).

In medical procedures, the RF energy used with this device, has been historically used in shrinking or removing soft-tissue, for surgical cutting, and for stopping bleeding. The device is cleared by the Food and Drug Administration (FDA) for use in coagulation (to assit with stoping bleeding and clotting of blood) of tissue within the digestive tract. The device has been used in areas outside the esophagus (inner lining of the throat), including the rectum to treat radiation proctitis. The stoppage of bleeding of radiation proctitis, using the HALO device, may be one method to control the bleeding.

The purpose of this study is to evaluate the effectiveness and record the results of treatment of radiation proctitis using the HALO device.

DETAILED DESCRIPTION:
This study is intended to prospectively gather information regarding the performance of an endoscope-mounted radiofrequency (RF) energy device, which utilizes RF energy for the coagulation of gastrointestinal tissue in the setting of bleeding of radiation proctitis. The study device, the HALO90 Ablation catheter, has an FDA 510(k) clearance for human use.

The study design is a single-site, prospective clinical trial to gather performance data regarding a 510(k)-cleared, endoscopically-guided radiofrequency energy ablation device for the coagulation of hemorrhagic radiation proctitis.

Study subjects will have experienced bloody stools due to proctitis following pelvic radiation for cancers of the prostate or uterine endometrium. The study will include female and male adult patients who have received pelvic radiotherapy for such indications as cancer of the prostate or endometrium and have subsequently experienced recurrent hemorrhagic radiation proctitis.

As part of this protocol, focal areas of the epithelial lining of the diseased colon, rectum, and/or anus will be treated with the study device. The aim is to obtain information about the hemostatic effect of this device. The treatment settings evaluated in this study have been previously established with this device in the esophagus in "treat and resect" protocols, as well as in clinical trials for Barrett's esophagus with long-term follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. History of pelvic irradiation. (Last radiation treatment must be greater than 6 months prior.)
2. Recurrent bloody stools.
3. Symptoms for > 3 months.
4. No active infection or ulceration.
5. Diagnosis of radiation proctitis by endoscopic criteria.
6. Other sources of bloody stools, such as colon cancer, ulcerative colitis, or hemorrhoids, have been ruled out by prior colonoscopy.
7. Age ≥ 18 years old.
8. Subject is able to tolerate endoscopy and sedation.
9. Subject agrees to participate, fully understands content of the informed consent, and signs the informed consent form (ICF).

Exclusion Criteria:

1. History of anal incontinence, rectal resection or anorectal malignancy.
2. Presence of anorectal fistulae or stenoses preventing passage of the endoscope and device.
3. Pregnancy and breastfeeding mothers
4. Subject is unable to provide informed consent for this study.
5. Pelvic irradiation within the last 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2008-07; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey M. Marks, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Case Medical Center, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ablation Catheter
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ablation Catheter
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 77
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: As this is a feasibility trial, the plan is to evaluate safety and efficacy in relation to adverse events in a small population (20 max) of patients.
Time Frame: 1 year
Population: There was no analysis of the data. Feasibility study with only one subject enrolled
Measure: Number; unit: partipants
Groups:
- Ablation Treatment: Subjects with radiation proctitis who met inclusion criteria
Arm/Group | Ablation Treatment
Number analyzed (Participants) | 1
partipants | 0

ADVERSE EVENTS:
Arm/Group | Ablation Catheter
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ablation Catheter (N=1)
Rectal Bleeding (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No